CLINICAL TRIAL: NCT06402357
Title: Salvage Focal Therapy Via High Intensity Focused Ultrasound (HIFU) in Radiorecurrent Localized Prostate Cancer
Brief Title: High Intensity Focused Ultrasound in Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: EDAP-TMS Focal One (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF-GU-009; IRB202401126 (Other: University of Florida)
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; high intensity focused ultrasound; focal therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- High Intensity Focused Ultrasound (Experimental)
  Interventions: Device: Focal One high intensity focused ultrasound device

INTERVENTIONS:
Device: Focal One high intensity focused ultrasound device — Participants will be treated with one session of high intensity focused ultrasound using the Focal One device.

SUMMARY:
This study will investigate the efficacy of focal high intensity focused ultrasound (HIFU) in patients with localized radiorecurrent prostate cancer. This study will also investigate the change in participant quality of life after HIFU therapy as compared to before HIFU therapy.

DETAILED DESCRIPTION:
Focal therapy is increasingly popular due to its minimal side effect profile. Furthermore, HIFU has demonstrated favorable oncologic outcomes in well selected patients, including those with intermediate and high risk disease. In patients with radiorecurrent prostate cancer there remains a paucity of data on the value of focal therapy. Review of focal HIFU rather than whole gland HIFU is based on largely retrospective data and in an era where mpMRI and PSMA PET was not yet widely implemented thus not reflecting the current patient population seeking this care. In fact, and to the investigators' knowledge, only one study has prospectively evaluated focal HIFU therapy in radiorecurrent prostate cancer. Further evaluation into the value of focal HIFU in select men with localized radiorecurrent clinically significant prostate cancer is needed (clinically significant prostate cancer defined as GG2 or above. GG1 prostate cancer will not be considered clinically significant prostate cancer), both in terms of oncologic and functional outcomes as this patient population is increasing.

ELIGIBILITY:
Inclusion Criteria:

* Patient has elected to undergo focal high intensity focused ultrasound therapy for radiorecurrent prostate cancer
* Males who are ≥ 18 years of age
* Eastern Cooperative Oncology Group Performance Status of 0-3
* A history of prostate cancer treated with radiation therapy +/- hormone therapy
* MRI or prostate-specific membrane antigen (PSMA) PET region of interest (ROI)
* Biopsy proven clinically significant prostate cancer (GG2 or above) recurrence within or ipsilateral to the ROI lesion (within 6 months of the MRI/PET).
* Contralateral grade group 1 (GG1) prostate cancer disease to the ROI
* PSMA PET negative for metastatic disease (within 6 months of the biopsy)
* Subjects must not have more than one active malignancy at the time of enrollment (Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen [as determined by the treating physician and approved by the PI] may be included).
* Written informed consent obtained from the subject and the subject agrees to comply with all the study-related procedures.

Exclusion Criteria:

* Contraindication to high intensity focused ultrasound (latex allergy, absent rectum, prior rectal fistula or significant rectal surgery making insertion of transrectal probe non-feasible or dangerous.)
* Hormone therapy within 6 months of the screening period (Hormone therapy includes oral (relugolix, abiraterone, enzalutamide, apalutamide, darolutamide, casodex) injections (firmagon, Lupron))
* History of Inflammatory Bowel Disease actively treated in last 3 years
* Evidence of ≥ cT3 recurrent disease on imaging
* Bilateral clinically significant prostate cancer
* Presence of brachytherapy seeds still implanted
* Presence of fiduciary markers which directly impede the successful treatment of the lesion of concern, as decided upon by the surgeon upon review of imaging
* Large Calcification on CT or transrectal ultrasound which, as per the review of the surgeon, limits or hinders a quality high intensity focused ultrasound to the region of interest
* Urethral stricture disease that has been active over the last 6 months or required further treatment than clean intermittent catheterization
* No prior radiation therapy for prostate cancer
* Subjects without a ROI on MRI or PET
* Metastatic disease or locally advanced disease (defined by pelvic lymph node involvement or T4 disease) on PSMA PET
* History of any other disease, metabolic dysfunction, clinical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician.
* Prisoners or subjects who are involuntarily incarcerated, or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
In-field failure-free survival | 12 months
  Evaluate the in-field failure-free survival (IFFFS) of localized radiorecurrent prostate cancer patients receiving focal HIFU treatment at 12 months. IFFFS is defined as the absence of biopsy proven clinically significant prostate cancer in the treated zone.

SECONDARY OUTCOMES:
Local failure-free survival | 12 months
  Evaluate the local failure-free survival (LFFS) of localized radiorecurrent prostate cancer patients receiving focal HIFU treatment at 12 months. LFFS is defined as the absence of biopsy proven clinically significant prostate cancer both in and out of the treated zone.
Complication rates | 12 months
  Determine the complication rates (Clavien Dindo >3) within the first 12 months. Complications include urinary tract infection, hematuria, urinary retention, stricture, bladder neck contracture, and incontinence.
Change in quality of life metrics | 6 months
  Determine the change from baseline in the International Prostate Symptom Score questionnaire total score at 6 months after HIFU treatment.
Change in quality of life metrics | 12 months
  Determine the change from baseline in the International Prostate Symptom Score questionnaire total score at 12 months after HIFU treatment.
Change in quality of life metrics | 6 months
  Determine the change from baseline in International Index of Erectile Function questionnaire scores at 6 months after HIFU treatment.
Change in quality of life metrics | 12 months
  Determine the change from baseline in International Index of Erectile Function questionnaire scores at 12 months after HIFU treatment.
Time from HIFU to whole gland or systemic therapy | 3 years
  Determine the time from HIFU to whole gland or systemic therapy
Time from HIFU to androgen deprivation therapy onset | 3 years
  Determine the time from HIFU to androgen deprivation therapy onset

CONTACTS AND LOCATIONS:
Overall Officials: Tarik Benidir, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States